CLINICAL TRIAL: NCT06312215
Title: Effect Of Open And Closed System Peripheral Catheters Used In Pediatric Services On Insertion Success, Duration Of Stay, And Development Of Complications: A Randomized Controlled Study
Brief Title: Effect Of Open And Closed System Peripheral Catheters Used In Pediatric Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Duygu Sonmez Duzkaya, Principal Investigator, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1763831
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Child, Only; Catheter Infection; Catheter Complications
Keywords: Closed System Peripheral Catheter; Peripheral Catheter; child

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed System Peripheral Catheters (Experimental): After the area where the catheter would be inserted was cleaned with an antiseptic solution and allowed to dry, a closed-system catheter was applied. Closed-system catheters are devices that allow access through needleless mechanisms, protecting the patient from accidental needle puncture injuries. They have mechanisms preventing blood leakage or pathogen entry.
  Interventions: Other: Closed-system catheter
- Control (No Intervention): After the area where the catheter would be inserted was cleaned with an antiseptic solution and allowed to dry, a catheter was applied.

INTERVENTIONS:
Other: Closed-system catheter — Closed-system catheters was applied
  Arms: Closed System Peripheral Catheters

SUMMARY:
The study was conducted as a randomized controlled experimental research to examine the effects of open and closed system peripheral catheters on the success of insertion, duration of stay, and development of complications in children aged 1-18 years in pediatric services. The population of the study consisted of children admitted to the Pediatric Services of the Istanbul Faculty of Medicine, and the sample included a total of N=80 children who met the sample criteria and underwent catheter insertion between May 2023 and October 2023. The sample was divided into two groups: closed system peripheral venous catheter group (n=40) and open system peripheral venous catheter group (n=40). The data of the study were collected using a Data Collection Form, Peripheral Venous Catheter Monitoring Form, Visual Infusion Phlebitis Detection Scale, and Pediatric Peripheral Intravenous Infiltration Scale

DETAILED DESCRIPTION:
The study was conducted as a randomized controlled experimental research to determine the impact of open and closed system peripheral catheters on the success of insertion, duration of stay, and the development of complications (infiltration, phlebitis) in children aged 1-18 years.

Location and Characteristics of the Study:

The research data were collected from pediatric patients in the Department of Pediatric Health and Diseases at Istanbul University Istanbul Faculty of Medicine. The pediatric services within the Department include Gastrohepatology, Neurology, Nutrition and Metabolism, Cardiology, Allergy and Immunology, Nephrology, Rheumatology, Endocrinology, and Chest Diseases, comprising a total of 47 service beds.

Study Population and Sample:

The study population consisted of children admitted to the pediatric services of Istanbul University Istanbul Faculty of Medicine between May 2023 and October 2023. The sample size was determined based on literature findings (Boztepe and Abusfia, 2015), considering a type I error rate of 0.05, a test power of 0.91 (α= 0.05, 1-β= 0.95). The minimum sample size for each group was calculated as 66 (n=33). However, to mitigate the possibility of losing cases, a total sample size of 80 patients was determined, with 40 patients in each group. Therefore, 40 patients would constitute the open system catheter group, and 40 patients would form the closed system catheter group. The selection of the sample was carried out through simple randomization based on predefined criteria for grouping the children.

Randomization:

In the study, there are two groups: the study group using closed system peripheral catheters and the control group receiving the routine procedure of the clinic with open system peripheral catheters. Children meeting the inclusion criteria were assigned to groups through a randomization process.

Subsequently, whenever a child meeting the inclusion criteria presented to the pediatric service, a nurse working in the unit, other than the researcher, asked the child to randomly select a piece of paper from a bag. If the paper indicated "control group," the child was assigned to the control group; if it indicated "study group," the child was assigned to the study group.

This randomization method, utilizing a simple and practical approach with the use of paper lots from a bag, ensures that each eligible child has an equal chance of being assigned to either the control or study group. The process helps minimize bias and ensures a more balanced distribution of characteristics across the groups, contributing to the reliability of the study results.

Data Collection:

In the pediatric service where the research was conducted, peripheral venous access and care for children were carried out by nurses using an open system catheter. The control group in this study consisted of the open system catheter group.

Data collection was performed in 6 stages:

Stage: Before the data collection process, a pilot application was conducted with 10 children to assess the suitability of the forms used in the research. Final adjustments were made to the forms after the pilot application.

Stage: Children included in the sample (aged 6 and older) and their parents were informed about the research, and verbal and written consents (informed consent) were obtained.

Stage: Patients meeting the sample selection criteria were randomly and equally distributed into two groups using the randomization method (1st group: control group with open system peripheral catheter application (n=40), 2nd group: study group with closed system peripheral catheter application (n=40)). It was ensured that the parents of children in both groups were present.

Stage: Before the procedure, the researcher filled out the "Patient Identification Form" for all children in the groups.

Stage: According to the group to which the child belonged, the researcher applied the "Peripheral Catheter Insertion and Removal Protocol." The protocol included the following steps:

Hands were washed, and necessary materials (gloves, cotton, an appropriately sized catheter for the child, 0.5% chlorhexidine-containing 70% alcohol, transparent drape, venous valve, saline solution, syringe) were prepared.

The area for catheter insertion was selected (upper extremity veins). Using aseptic technique, the catheter was inserted using the appropriate method (gloves were worn, the catheter area was wiped three times with a solution of 2% chlorhexidine-containing 70% alcohol, and it was allowed to dry; the cleaned area was not touched after wiping).

After inserting the catheter, it was secured using a transparent drape for easy observation.

For children with open system peripheral catheters, a venous valve was attached after catheter insertion to reduce movement of the catheter.

Catheter dressing was changed if there was moisture, looseness, or noticeable contamination.

Stage: After the insertion of the peripheral venous catheter (PVC), children were monitored daily using the "Daily Monitoring Form" until 48 hours after removal.

Data Analysis:

The data obtained in the research were analyzed using the Statistical Package for Social Sciences (SPSS) 22.0 program. Normal distribution analysis was conducted, and it was determined that the data did not follow a normal distribution. Therefore, non-parametric tests were employed for the analyses.

For qualitative variables, frequency and percentage calculations were performed.

For quantitative variables, mean, standard deviation, and median tests were conducted.

Categorical variables were compared using the Chi-square test, while quantitative variables were compared using the Mann-Whitney U test.

A significance level of p<0.05 was considered in the analyses. This means that statistically significant differences were considered when the p-value was below 0.05. This value represents the significance level used to determine differences between various groups in the study.

ELIGIBILITY:
Inclusion Criteria:

* • Being between 1 and 18 years of age,

  * Having a catheter requirement for at least 72 hours,
  * The catheter being inserted in the admitting service,
  * Catheters not being inserted under emergency conditions,
  * Absence of other catheters (central venous, arterial, PICC line, etc.),
  * Body temperature not exceeding 38°C,
  * Absence of skin issues in the catheter area,
  * Not undergoing chemotherapy treatment,
  * The catheter being inserted in the upper extremity,
  * Willingness to voluntarily participate in the study.

Exclusion Criteria:

* Being under 1 year of age or over 18 years,
* Having a catheter requirement of less than 72 hours,
* Peripheral catheters being inserted under emergency conditions,
* Presence of other catheters in the child (central venous, arterial, PICC line, etc.),
* Body temperature exceeding 38°C,
* Presence of skin issues in the area where the catheter will be inserted,
* Undergoing chemotherapy treatment,
* Unwillingness to voluntarily participate in the study.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Patient Identification Form | 1 day
  he Patient Identification Form has been prepared by reviewing relevant literature. It consists of 27 questions, encompassing patient-specific information and catheter characteristics.
Daily Monitoring Form | 1 day
  his form, comprised of 8 questions, has been designed to monitor patients on a daily basis, covering aspects such as catheter day, fluids administered, phlebitis score, infiltration score, skin characteristics, and signs of infection. Nurses used the Daily Monitoring Form to observe and record patient conditions on a daily basis.
Visual Infusion Phlebitis Assessment Scale, Staging Key - Peripheral IV'sVIPAS | 1 day
  Developed by Alyce Schultze and Paulette Gallant, this scale was published by the Infusion Nurses Society in 2011 for the purpose of grading phlebitis. The scale involves observing the possible risks of the catheter during the administration of treatment through a peripheral intravenous catheter. It also includes grading the symptoms of phlebitis at each stage if phlebitis develops. The content validity index value of the scale was found to be 0.97
Pediatric peripheral intravenous infiltration assessment tool | 1 day
  Pediatric peripheral intravenous infiltration assessment tool: Developed by Simona and evaluated for its psychometric properties, the Pediatric Peripheral Intravenous Infiltration Scale has undergone Turkish validity and reliability assessments by Temizsoy et al. (2017) and is suitable for use in newborns. Cohen kappa value of the scale was 0.80 (p<0.001) and Pearson correlation coefficient was r=0.95 (p<0.001). The Cronbach's alpha coefficient of the scale is 0.966, which shows that the level of infitration increases as the stages increase in the evaluation made in five stages.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Mersin, Turkey (Türkiye)

REFERENCES:
- [Background] Amjad I, Murphy T, Nylander-Housholder L, Ranft A. A new approach to management of intravenous infiltration in pediatric patients: pathophysiology, classification, and treatment. J Infus Nurs. 2011 Jul-Aug;34(4):242-9. doi: 10.1097/NAN.0b013e31821da1b3. PMID 21734520
- [Background] Clark E, Giambra BK, Hingl J, Doellman D, Tofani B, Johnson N. Reducing risk of harm from extravasation: a 3-tiered evidence-based list of pediatric peripheral intravenous infusates. J Infus Nurs. 2013 Jan-Feb;36(1):37-45. doi: 10.1097/NAN.0b013e3182798844. PMID 23271150
- [Background] Corley A, Ullman AJ, Mihala G, Ray-Barruel G, Alexandrou E, Rickard CM. Peripheral intravenous catheter dressing and securement practice is associated with site complications and suboptimal dressing integrity: A secondary analysis of 40,637 catheters. Int J Nurs Stud. 2019 Dec;100:103409. doi: 10.1016/j.ijnurstu.2019.103409. Epub 2019 Aug 28. PMID 31629208
- [Background] Doellman D, Hadaway L, Bowe-Geddes LA, Franklin M, LeDonne J, Papke-O'Donnell L, Pettit J, Schulmeister L, Stranz M. Infiltration and extravasation: update on prevention and management. J Infus Nurs. 2009 Jul-Aug;32(4):203-11. doi: 10.1097/NAN.0b013e3181aac042. PMID 19605999
- [Background] Duncan M, Warden P, Bernatchez SF, Morse D, (2018), A bundled approach to decrease the rate of primary bloodstream infections related to peripheral intravenous catheters, J Assoc Vasc Access, 23(1), 15-22.
- [Background] Arias-Fernandez L, Suerez-Mier B, Martinez-Ortega MD, Lana A. Incidence and risk factors of phlebitis associated to peripheral intravenous catheters. Enferm Clin. 2017 Mar-Apr;27(2):79-86. doi: 10.1016/j.enfcli.2016.07.008. Epub 2016 Sep 16. English, Spanish. PMID 27640931
- [Background] Gonzalez Lopez JL, Arribi Vilela A, Fernandez del Palacio E, Olivares Corral J, Benedicto Marti C, Herrera Portal P. Indwell times, complications and costs of open vs closed safety peripheral intravenous catheters: a randomized study. J Hosp Infect. 2014 Feb;86(2):117-26. doi: 10.1016/j.jhin.2013.10.008. Epub 2013 Dec 1. PMID 24373830
- [Background] Gorski LA, Hadaway L, Hagle ME, Broadhurst D, Clare S, Kleidon T, Meyer BM, Nickel B, Rowley S, Sharpe E, Alexander M. Infusion Therapy Standards of Practice, 8th Edition. J Infus Nurs. 2021 Jan-Feb 01;44(1S Suppl 1):S1-S224. doi: 10.1097/NAN.0000000000000396. No abstract available. PMID 33394637